CLINICAL TRIAL: NCT05236374
Title: Effects of Daily Beef Intake, as a Component of a Heart-Healthy Diet, on Cellular Zinc Status and Vascular Function in Older Adults
Brief Title: Effects of Daily Beef Intake, as a Component of a Heart-Healthy Diet on Cellular Zinc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1806393
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Zinc Deficiency; Inflammation; Metabolic Diseases; Vascular Diseases
MeSH Terms: conditions — Inflammation; Metabolic Diseases; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Crossover comparison of a mixed diet including green leafy vegetables, fruits, whole grains, seeds, and nuts; with beef versus non-meat sources of additional protein and zinc, over two 4-week metabolic study periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beef Protein (Experimental): A beef stew, providing 8.8 mg zinc, 37.9 mg protein (approximately 500 kcal/d energy);
  Interventions: Other: Beef protein
- Animal Protein (Active Comparator): A control plant protein stew, providing 8.8 mg zinc, 37.9 mg protein (approximately 500 kcal/d energy);
  Interventions: Other: Beef protein

INTERVENTIONS:
Other: Beef protein — Animal protein source

SUMMARY:
The objective of the current study is to test the overarching hypothesis that the beef nutritive matrix is uniquely suited to direct dietary zinc to cellular compartments for improved metabolic function, leading to a greater effect on health outcomes. Specifically, whether beef, as a component of a healthy meal, will promote the absorption of zinc into cells, where the zinc will have greater effects on zinc-dependent metabolic processes supporting cardiovascular health. To maximize the observability of these beef-related effects, individuals who are 55- to 70-year-old who generally have a higher risk of zinc deficiency and cardiovascular disease will be enrolled.

DETAILED DESCRIPTION:
This study will examine whether daily beef intake will promote the absorption of dietary zinc into cells, leading to improved cellular zinc status and microvascular function. The study design will be a crossover comparison of a mixed diet including green leafy vegetables, fruits, whole grains, seeds, and nuts; with beef versus non-meat sources of additional protein and zinc, over two 4-week metabolic study periods.

Outcomes will include cellular zinc status determined by erythrocyte zinc tracer exchange (primary), and microvascular function expressed as reactive hyperemia index (RHI). Previous studies have demonstrated that zinc tracer exchange with red blood cells (RBC) is highly sensitive to changes in zinc nutriture. Thus, cellular zinc status will be determined using a novel and cost-effective adaptation of this approach, modeling zinc tracer exchange with freshly-sampled RBC. As intracellular zinc can regulate vascular tone, microvascular function will be measured, using digital peripheral tonometry, will be used as a functional index of both cellular zinc status and vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal female 55-70 years of age
* Women: lack of menses for at least two years.
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* Self-reported stable dose of prescribed medications for a minimum of 6 months
* BMI 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Prescribed metaformin, statins or medications known to interfere with zinc, protein, or lipid metabolism
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet (e.g. Adkins, Keto, Paleo, etc.)
* Fruit consumption ≥ 3 cups/day
* Regular consumption of strawberries (2-3 servings/week)
* Vegetable consumption ≥ 4 cups/day
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Alcohol intake greater than 2 drinks in a day for men, or 1 drink in a day for women.
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Peripheral artery disease Raynaud's syndrome or disease
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Unwillingness to stop any supplement use six weeks prior to study initiation, including multivitamin/mineral, powders, herbal, plant or botanical, pro- and prebiotics, and oil supplements.
* Smoking, vaping, cannabis use
* Current enrollee in a clinical research study.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
microvascular function | 4 weeks
  microvascular function as measured by digital tonometry (EndoPAT2000)
intracellular zinc status | 4 weeks
  intracellular zinc status determined by erythrocyte zinc tracer exchange

SECONDARY OUTCOMES:
plasma lipids | 4 weeks
  Circulating level of total cholesterol, triglycerides, HDL cholesterol, non-HDL cholesterol, with LDL cholesterol (calculated)
plasma fatty acids | 4 weeks
  Circulating levels of non-esterified fatty acids
plasma oxylipins | 4 weeks
  enzyme and non-enzyme derived non-esterified fatty acid metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — Distinguished Professor Emeritus of Nutrition
Locations (1):
- University of California, Davis; Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No